CLINICAL TRIAL: NCT07273513
Title: "Smart Family Doctor" Assisted Comprehensive Management of Secondary Prevention Among Post Revascularization Patients
Acronym: SMART II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Xin Yuan, Professor, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FW-YX-002
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hypertension; Diabete Mellitus; Hyperlipidemia; Post PCI; Post CABG
Keywords: smartphone; AI-assisted; Revascularization management; metabolic management; Smart family doctor
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: The intervention in this study is the implementation of the 'Smart family doctor' system, a digital health management tool designed to support secondary prevention in post-CABG patients. This system leverages knowledge from coronary artery disease (CAD) secondary prevention guidelines, expert consensus, and a knowledge base addressing common post-revascularization issues. It is powered by a large-scale, medical knowledge-enhanced conversational model, enabling personalized interactions with patients to guide their recovery and lifestyle management following surgery.
Masking Description: Data manager and statistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- "Smart family doctor" assisted management (Experimental): "Smart family doctor", an AI-assisted applications with personalized interactions in 24 hours and 7 days a week.
  Interventions: Behavioral: Smart family doctor
- Health managers (Experimental): 3-hour health management guidance from a health manager once a week.
  Interventions: Behavioral: Health manager
- Usual care (Placebo Comparator): Usual post-surgery management
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Smart family doctor — Participants will be provided "Smart family doctor", which is an AI-assisted applications with personalized interactions. The content includes, but is not limited to: (1) General educational content, covering basic health knowledge on diseases, risk factors, and treatment methods; (2) Targeted health information, such as more specific guidance on blood pressure and blood sugar control, medication adherence, exercise, and smoking cessation; (3) Personalized disease management guidance, providing tailored reminders for patients regarding medication, diet, exercise, and medical visits. Patients can also directly report their latest self-measured blood pressure, blood lipid, blood sugar levels, and medication adherence to receive treatment and medication guidance from the 'Smart family doctor'.
  Arms: "Smart family doctor" assisted management
Behavioral: Health manager — Participants will received 3-hour health management guidance from a health manager once a week, including guidance on healthy lifestyle, medication treatment, and rehabilitation advice.
  Arms: Health managers
Behavioral: Usual Care — Participants will receive usual secondary prevention management.
  Arms: Usual care

SUMMARY:
This study aims to evaluate the effect of an AI-assisted "Smart family doctor" digital health management tool on improving the control rates of hypertension, diabetes, and dyslipidemia in post-revascularization patients. A randomized controlled trial design will be used, involving approximately 10-20 hospitals and 951 participants. Eligible participants are adults aged between 18 and 80 years, post-CABG or post-PCI patients with hypertension, diabetes, and dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years.
* Underwent CABG or PCI more than 3 months prior and have concurrent hypertension, diabetes, and dyslipidemia.
* At least one of the following criteria is meet:
* Systolic blood pressure no less than 130 mmHg or diastolic blood pressure no less than 80 mmHg
* HbA1c no less than 7%
* LDL-C no less than 1.4 mmol/L
* Signed informed consent.

Exclusion Criteria:

* History of heart failure or severe arrhythmias.
* Presence of other severe underlying conditions such as cancer or liver and kidney insufficiency.
* Pregnancy, lactation, or plans for pregnancy within the next year.
* Cognitive, communication impairments, or limitations in daily activities.
* Unable to use smartphone.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 951 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
The control rates of hypertension, diabetes and hyperlipidemia | 6-month
  All cretria are meet: 1) Systolic blood pressure less than 130 mmHg and diastolic blood pressure less than 80 mmHg. 2) HbA1c less than 7%. 3) LDL-C less than 1.4 mmol/L.

SECONDARY OUTCOMES:
Blood Pressure Control Rate | 6-month
  The proportion of patients with systolic blood pressure less than 130 mmHg and diastolic blood pressure less than 80 mmHg.
Blood glucose Control Rate | 6-month
  The proportion of patients with HbA1c less than 7%.
Blood lipid Control Rate | 6-month
  The proportion of patients with LDL-C less than 1.4mmol/L.
Systolic blood pressure | 6-month
  Systolic blood pressure measured at the local site.
Diastolic blood pressure | 6-month
  Diastolic blood pressure measured at the local site.
Fasting blood glucose | 6-month
  Fasting blood glucose analyzed at central lab.
HbA1c | 6-month
  HbA1c analyzed at central lab.
Total cholesterol | 6-month
  Total cholesterol analyzed at central lab.
LDL-C | 6-month
  LDL-C analyzed at central lab.
HDL-C | 6-month
  HDL-C analyzed at central lab.
Triglycerides | 6-month
  Triglycerides analyzed at central lab.
Medication adherence (4-item Morisky Medication-Taking Adherence Scale) | 6-month
  Medication adherence measured by MMAS-4. The score range from 0 to 4. The higher score indicated the better medication adherence.
Coronary artery disease-related quality of life (the Seattle Angina Questionnaire) | 6-month
  Coronary artery disease-related quality of life assessed with the Seattle Angina Questionnaire (SAQ). The score range from 0 to 100. The higher score indicated the better coronary artery disease-related quality of life.
Smoking Rate | 6-month
  The proportion of patients who have smoked within the past month.

OTHER OUTCOMES:
Major adverse cardiovascular events (MACE) | 6-month
  The composite endpoint of cardiovascular death, myocardial infarction, stroke, or hospitalization due to cardiovascular disease.
BMI | 6-month
  Body mass index (BMI) is calculated as weights (kg) divided by the square of heights (meters).
Waist circumference | 6-month
  Waist circumference is measured at local site.
Rehospitalization rate | 6-month
  The proportion of patients who had hospitalization
The number of emergency visit | 6-month
  The number of emergency visit during follow-up period
System usability (system usability scale) | 6-month
  System usability measured by system usability scale. The proportion of patients who scaled system usability more than 68 points.
Subgroup-age | 6-month
  Primary outcome analyses in age subgroups: <=65, >65 years
Subgroup-sex | 6-month
  Primary outcome analyses in sex subgroups: women, men
Subgroup-education level | 6-month
  Primary outcome analyses in education level subgroups: less than high school, high school or higher
Subgroup-smoking status | 6-month
  Primary outcome analyses in smoking status subgroups: current smoking, no smoking
Subgroup-baseline BP level | 6-month
  Primary outcome analyses in baseline BP level subgroups: SBP/DBP>=130/80 mmHg, <130/80 mmHg
Subgroup-baseline LDL-C level | 6-month
  Primary outcome analyses in baseline LDL-C level subgroups: <1.4 mmolL, >=1.4 mmol/L
Subgroup-baseline HbA1c level | 6-month
  Primary outcome analyses in baseline HbA1c level subgroups: <7%, >=7%

CONTACTS AND LOCATIONS:
Overall Officials: Xin Yuan, PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data that support the findings of this study are available from the corresponding author, upon reasonable request, only for authorized research. Their use is subjected to an agreement with the promotor (Fuwai Hospital) and the principal investigator (Dr Xin Yuan) of the SMART II study. Pseudonymised data that support the findings of this study are available from the promotor (Fuwai Hospital) upon reasonable request, subject to a specific agreement with the promotor (involving the principal investigator) and subject to regulatory proceedings due to data protection applicable laws. Access conditions are to be determined depending on the nature of the request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the end of the study
Access Criteria: Anonymized data that support the findings of this study are available from the corresponding author, upon reasonable request, only for authorized research. Their use is subjected to an agreement with the promotor (Fuwai Hospital) and the principal investigator (Dr Xin Yuan) of the SMART II study. Pseudonymised data that support the findings of this study are available from the promotor (Fuwai Hospital) upon reasonable request, subject to a specific agreement with the promotor (involving the principal investigator) and subject to regulatory proceedings due to data protection applicable laws. Access conditions are to be determined depending on the nature of the request.